CLINICAL TRIAL: NCT04183972
Title: Identification of Interscalene Brachial Plexus Automatically on Ultrasonography Using a Deep Neural Network
Brief Title: Identification of Interscalene Brachial Plexus on Ultrasonography Using a Deep Neural Network
Acronym: IBRUNNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yang, MD, Principal Investigator, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2019-502
Record Dates: First submitted 2019-11-19; First posted 2019-12-03 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Ultrasound Therapy; Complications
Keywords: peripheral nerve block; ultrasound image; deep neural network; brachial plexus

STUDY DESIGN:
Intervention Model Description: Patients who have been scheduled to surgery will be recruited for collecting ultrasound images.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image collecting Group (Experimental): An computer algorithm will be developed and evaluated by these image data.
  Interventions: Procedure: ultrasound examination

INTERVENTIONS:
Procedure: ultrasound examination — the participants will be placed in the supine position, with head turned slightly away from the operating side and arms beside the body. The operator will identify right and left interscalene brachial plexuses by ultrasound equipment (Sonosite EDGE or GE LOGIQ e). Clear images and videos of brachial plexus will be captured and saved.

SUMMARY:
The purpose of the study is to develop and validate an algorithm based on deep neural networks (DNNs) to identify interscalene brachial plexus on ultrasonography automatically.

DETAILED DESCRIPTION:
The investigators plan to develop a deep learning-based network to automatically identify interscalene brachial nerves on ultrasound images. The trained model will be validated on an independent dataset. The performance of the network will also be compared against practicing anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I or II
* scheduled for elective surgery

Exclusion Criteria:

* skin lesion or infection of neck
* any known peripheral neuropathy
* brachial nerve plexus injury
* previous injury or operation on neck
* pregnancy
* allergic to ultrasound gel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1126 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
The distance of the lateral midpoints of the nerve sheath contours | immediately after the procedure
  between model predictions and the ground truth; between nonexpert anesthesiologist predictions and the ground truth

SECONDARY OUTCOMES:
Accuracy, Sensitivity and specificity | immediately after the procedure
  Accuracy, Sensitivity and specificity of the network and nonexpert anesthesiologists
The percentage of the intersection over union | immediately after the procedure
  between model predictions and the ground truth; between nonexpert anesthesiologist predictions and the ground truth

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Yang, MD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang XY, Wang LT, Li GD, Yu ZK, Li DL, Guan QL, Zhang QR, Guo T, Wang HL, Wang YW. Artificial intelligence using deep neural network learning for automatic location of the interscalene brachial plexus in ultrasound images. Eur J Anaesthesiol. 2022 Sep 1;39(9):758-765. doi: 10.1097/EJA.0000000000001720. Epub 2022 Jul 20. PMID 35919026